CLINICAL TRIAL: NCT03247699
Title: Pharmacokinetics of the Basel Phenotyping Cocktail Combination Capsule
Acronym: CombiCapsIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2016-01766
Record Dates: First submitted 2017-08-04; First posted 2017-08-14 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: CYP450 Phenotyping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Basel phenotyping cocktail" capsule (Other)
  Interventions: Other: "Basel phenotyping cocktail" capsule
- "Basel phenotyping cocktail" individual components (Other)
  Interventions: Other: "Basel phenotyping cocktail" individual components

INTERVENTIONS:
Other: "Basel phenotyping cocktail" capsule — Oral intake of "Basel phenotyping cocktail" capsule and pharmacokinetics (PK) sampling
  Arms: "Basel phenotyping cocktail" capsule
Other: "Basel phenotyping cocktail" individual components — Oral intake of "Basel phenotyping cocktail" individual components and PK sampling
  Arms: "Basel phenotyping cocktail" individual components

SUMMARY:
Healthy Subjects will receive treatment orally with 120-200ml tap water in fasted state.

Treatment in period A is the "Basel phenotyping cocktail" capsule. Treatment in period B consists of simultaneous intake of isolated formulations. In both study arms peripheral venous and capillary blood (DBS) samples will be drawn

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years old
* Caucasian male volunteers
* Body mass index (BMI)18-30kg/m2,weight more than 50kg
* Full mental and legal capacity
* Signed informed consent prior to any study related procedure
* Ability to communicate in German or English, sufficient to comprehend and adhere to study protocol
* Systolic blood pressure (SBP) 100-145mmHg, diastolic blood pressure (DBP) 50-90mmHg and heart rate (HR) 45-90bpm (inclusive), measured on the leading arm*, after 5min in the supine position at screening Normal physical examination, vital signs, laboratory workup, and electrocardiogram (ECG)
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent at screening
* No other conditions or circumstances that might interfere with compliance with study protocol

Exclusion Criteria:

* Known hypersensitivity to any excipients of the drug formulations.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs, or which might increase the risk for toxicity.
* History or presence of smoking (within the last 3months prior to screening) or alcohol or drug abuse
* Intake of prescribed or otc medications, herbal preparations, and / or vitamin/dietary supplements within 2weeks prior to the intended start of study.
* Excessive caffeine consumption, defined as >800 mg per day at Screening Intake of food products (immediately before or during study) known to be inducers or inhibitors of CYP450

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-30 (Actual)

PRIMARY OUTCOMES:
Concentration-time profile in plasma | -5 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours
  Concentration-time Profiles assessed in Plasma over several time points measuring parent compounds and corresponding metabolites to calculate metabolic ratios
Concentration-time profile in capillary blood | -5 minutes, 5 minutes, 15 minutes, 30 minutes, 45 minutes, 60 minutes, 2 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours
  Concentration-time Profile assessed in capillary blood over several time points measuring parent compounds and corresponding metabolites to calculate metabolic ratios

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Krähenbühl, MD PhD, Principal Investigator — Universitätsspital Basel, Switzerland
Locations (1):
- Ambulantes Studienzentrum, Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
Results of Trial will be published in a peer reviewed Journal